CLINICAL TRIAL: NCT06807905
Title: Prospective, Interventional Study to Iivestigate the Efficiency and Biocompatibility in Hemodiafiltration Procedure
Brief Title: Efficiency and Biocompatibility in Hemodiafiltration Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Milena Andonova, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HDFCOMP
Record Dates: First submitted 2020-01-19; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: End Stage Renal Disease on Dialysis; Biocompatibility; Anticoagulation; Hemodiafiltration
Keywords: Dialysis; Hemodifiltraton; Biocompatibility; Anticoagulation; regional citrate anticoagulation; heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heparin anticoagulation (Active Comparator): Heparin anticoagulation in hemodiafiltration procedure
  Interventions: Drug: Heparin anticoagulation
- Citrate anticoagulation (Experimental): Hemodiafiltration will be performed with regional citrate anticoagulation
  Interventions: Drug: Citrate anticoagulation

INTERVENTIONS:
Drug: Heparin anticoagulation — Hemodiafiltration will be performed with heparine anticoagulation
  Arms: Heparin anticoagulation
Drug: Citrate anticoagulation — Patient will perform dialysis with citrate anticoagulation
  Arms: Citrate anticoagulation

SUMMARY:
Hemodiafiltration is a modern, increasingly used special hemodialysis method. Compared to hemodialysis, it allows greater clearance of medium- and high-molecular-weight molecules. Modern hemofiltration membranes are approaching the properties of the glomerular membrane in their properties.

During hemodiafiltration, blood contact with the semipermeable membrane and blood lines causes activation of the coagulation system, so anticoagulation during the procedure is absolutely necessary. Heparin is routinely used as a method of anticoagulation in hemodiafiltration. Regional citrate anticoagulation is used primarily in patients with risk of bleeding.

The purpose of our study is to evaluate the kinetics of citrate, calcium, and magnesium during hemodiafiltration and citrate anticoagulation, and in these way optimizing the citrate anticoagulation protocol during hemodiafiltration, and to compare the clearance of small and medium molecules between the two anticoagulations (citrate and heparin). The purpose of the study is also to compare biocompatibility parameters for heparin and citrate anticoagulation in hemodiafiltration.

DETAILED DESCRIPTION:
Aim of the study

Hemodiafiltration is a modern, increasingly used special hemodialysis method. Compared to hemodialysis, it allows greater clearance of medium- and high-molecular-weight molecules. Modern hemofiltration membranes are approaching the properties of the glomerular membrane in their properties.

During hemodiafiltration, blood contact with the semipermeable membrane and blood lines causes activation of the coagulation system, so anticoagulation during the procedure is absolutely necessary. Heparin is routinely used as a method of anticoagulation in hemodiafiltration. Regional citrate anticoagulation is used primarily in patients with risk of bleeding.

The purpose of our study is to evaluate the kinetics of citrate, calcium, and magnesium during hemodiafiltration and citrate anticoagulation, and in these way optimizing the citrate anticoagulation protocol during hemodiafiltration, and to compare the clearance of small and medium molecules between the two anticoagulations (citrate and heparin). The purpose of the study is also to compare biocompatibility parameters for heparin and citrate anticoagulation in hemodiafiltration.

Hypothesis

In the research, there are two hypotheses:

1. The removal of small and medium molecules is better at citrate than heparin hemodiafiltration.
2. The biocompatibility of the procedure is better with citrate than with heparin hemodiafiltration.

Backgorund

The hemodiafiltration procedure better removal of medium molecules compared to hemodialysis procedure. No comparisons were made in the literature for the removal of these molecules by heparin and citrate hemodiafiltration. Research has shown that citrate anticoagulation improves the biocompatibility of the dialysis system in hemodialysis, since many blood-body interactions with foreign substances are largely dependent on calcium and magnesium. Hemodiafiltration has not yet examined the biocompatibility of hemodiafiltration procedures with heparin or. citrate as an anticoagulant. In hemodiafiltration, the kinetics of citrate, calcium, and magnesium are unpredictable, since part of the calcium is also eliminated at the expense of the infusion, respectively. hemofiltration. Patients should be temporarily transferred to conventional hemodialysis if citrate anticoagulation is required. Given that we do not have this information so far, we will optimize the citrate anticoagulation protocol using this research.

Study design, method description, subjects

We will include 20 adult dialysis-dependent patients with end-stage renal impairment who are enrolled in a regular dialysis replacement dialysis program. In the study, patients will be randomized to two groups after obtaining written consent, which will differ in the order of anticoagulation used: 1) heparin anticoagulation group and then citrate anticoagulation, 2) citrate anticoagulation group and then heparin anticoagulation. Each patient will undergo two hemodiafiltration procedures, which will be study (research), one with heparin and one with citrate as an anticoagulant, so that each patient will be in control of himself. The first group of patients will use standard heparin. In the group of patients with citrate anticoagulation, the following protocol will be used: anticoagulation with 8% 3-sodium citrate, with a blood flow of 300 ml / min, with a dialysate flow of 500 ml / min. At the venous limb of the system, 1M CaCl2 will be added at an initial dose of 16-18 ml / h, which will then be adjusted according to the normal values of ionized calcium according to regular controls during the procedure (normal values of ionized calcium from 1.1-1.2 mmol / L). For the appropriate effect of anticoagulation, the value of ionized calcium in the dialysis circuit would be below 0.40 mmol / L (sampling point directly behind the filter). In both patient groups, gas analysis of venous blood, electrolytes (including magnesium, calcium and phosphorus), uremic toxins (urea, creatinine), B2-microglobulin will be monitored before and after the procedure. In the citrate group, the values of ionized calcium (before and after the filter) will be monitored at regular intervals during hemodiafiltration. We will also calculate the screening coefficient (SC) after 15 min. and just before the end of the procedure ( SC = 2D / (A+V), A = concentration on arterial line, V = concentration on venous line: D = concentration in filtrate or dialysate). The following biocompatibility parameters will be measured: hemogram (e. Leukopenia, thrombocytopenia), complement activation by C5a determination. Biocompatibility parameters will be measured before hemodiafiltration, after 15 min, after 1 hour, and after the end of the procedure. All dialysate will be collected, which is otherwise dumped into the water drain during routine work. Phosphate, B2-microglobulin, will be determined from all dialysate. The main outcome of the study is the screening coefficient for beta 2-microglobulin, the screening coefficient for phosphate is a secondary outcome.

Following the completion of the hemodiafiltration procedure, five patients in both groups will be subjected to electron microscopy after dialysis to evaluate cell adsorption, protein and clot formation on the dialysis membrane.

Expected results

We expect better removal efficiency of small and medium molecules in hemodiafiltration with citrate anticoagulation compared to standard heparin anticoagulation. With citrate anticoagulation, reduced activation of complement and hemostasis, leukocytes and platelets is expected. The results of the study will help to clarify the role of citrate anticoagulation in improving the biocompatibility of hemodiafiltration. With positive results, citrate anticoagulation during hemodiafiltration could be performed in all chronic dialysis patients in the future. We also expect better removal of low and medium molecular weight solutes in citrate anticoagulation, due to globally better anticoagulation and, consequently, better preservation of the permeability of the dialyzer membrane throughout the dialysis procedure.

ELIGIBILITY:
Inclusion Criteria:

* CKD on dialysis

Exclusion Criteria:

* AKI on dialysis
* patients on anticoagulant therapy
* systemic bacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
removal of small and medium molecules | during 4 hour dialysis
  The removal of small and medium molecules is different comparing citrate and heparin anticoagulation.

SECONDARY OUTCOMES:
biocompatibility | during 4 hour dialysis
  The biocompatibility of the procedure is different comparing citrate than with heparin anticoagulation.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Andonova, MD, Principal Investigator — University Medical Centre Ljubljana, Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes